CLINICAL TRIAL: NCT02224729
Title: Phase II Study of Bendamustine, Bortezomib, and Dexamethasone (BBD) for Newly Diagnosed Patients With Multiple Myeloma
Brief Title: Bendamustine Hydrochloride, Bortezomib, and Dexamethasone in Treating Patients With Newly Diagnosed Multiple Myeloma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Cancer Center at Thomas Jefferson University (Other)
Responsible Party: Sponsor
Organization: Thomas Jefferson University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14D.300; 2014-025 (Other: CCRRC); JT 6192 (Other: JeffTrial Number)
Record Dates: First submitted 2014-08-21; First posted 2014-08-25 (Estimated); Results first posted 2018-06-07 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Stage I Multiple Myeloma; Stage II Multiple Myeloma; Stage III Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Bendamustine Hydrochloride; Bortezomib; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Bendamustine, Bortezomib, Dexamethasone (Standard) (Experimental): Patients receive bendamustine hydrochloride IV over 30 minutes on days 1 and 2; bortezomib SC on days 1, 8, 15, and 22; and dexamethasone PO on days 1, 8, 15, and 22. Treatment repeats every 35 days for 4 courses in the absence of disease progression or unacceptable toxicity. Patients achieving less than a VGPR or with more than 10% bone marrow plasmacytosis may receive 2 additional courses.
  Interventions: Drug: Bendamustine hydrochloride; Drug: Bortezomib; Drug: Dexamethasone

INTERVENTIONS:
Drug: Bendamustine hydrochloride — Given IV
  Other Names: Treakisym; Ribomustin; Levact; Treanda; SDX-105
Drug: Bortezomib — Given SC
  Other Names: PS-341; Velcade; Cytomib
Drug: Dexamethasone — Given PO

SUMMARY:
This phase II trial studies side effects and how well bendamustine hydrochloride, bortezomib, and dexamethasone work in treating patients with newly diagnosed multiple myeloma. Drugs used in chemotherapy, such as bendamustine hydrochloride and dexamethasone, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Bortezomib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Giving bendamustine hydrochloride with bortezomib and dexamethasone may kill more cancer cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Establish the response rate of induction therapy following 4 cycles of the combination regimen bendamustine (bendamustine hydrochloride), bortezomib and dexamethasone (BBd) in patients with newly diagnosed multiple myeloma.

II. Describe the tolerability and toxicities of this regimen. III. Provide one-year progression-free survival and one-year overall survival data following this therapeutic strategy.

OUTLINE:

Patients receive bendamustine hydrochloride intravenously (IV) over 30 minutes on days 1 and 2; bortezomib subcutaneously (SC) on days 1, 8, 15, and 22; and dexamethasone orally (PO) on days 1, 8, 15, and 22. Treatment repeats every 35 days for 4 courses in the absence of disease progression or unacceptable toxicity. Patients achieving less than a very good partial response (VGPR) or with more than 10% bone marrow plasmacytosis may receive 2 additional courses.

NOTE: Patients requiring immediate reduction in paraprotein during course 1 only receive bendamustine hydrochloride IV over 30 minutes on days 1 and 2; bortezomib IV on days 1, 4, 8, and 11; and dexamethasone PO on days 1-4.

After completion of study treatment, patients are followed up for 1 year.

ELIGIBILITY:
Inclusion Criteria:

1. New diagnosis of multiple myeloma with no prior history of systemic treatment (Exceptions include corticosteroids, bisphosphonates, single agent cyclophosphamide, <= 21 days of the first cycle of a planned regimen
2. >= 18 years of age
3. ECOG <= 3
4. Signed informed consent
5. Measurable serum paraprotein on SPEP or serum free light chains and ratio, or quantifiable Bence-Jones proteinuria on 24 hour urine specimen. If the monoclonal protein has merged with the beta region we will follow the serum immunoglobulin of the involved heavy chain and comment on either partial remission (PR, as judged by two protocol investigators) or complete remission (CR, as defined by the achievement of PR as above and the resolution of the monoclonal protein by immunofixation in the serum and urine.)

Exclusion Criteria:

1. Failure to sign informed consent
2. Smoldering myeloma, monoclonal gammopathy of undetermined significance (MGUS), or plasma cell leukemia
3. History of previously treated smoldering myeloma
4. Grade 3 or above peripheral neuropathy
5. Uncontrolled human immunodeficiency virus (HIV)
6. Active hepatitis A, B or C
7. Pregnant or lactating females
8. Total bilirubin >3 times the upper limit of normal
9. ASLT/ALT > 2.5 times the upper limit of normal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2014-08-25 (Actual); Primary Completion 2016-04-21 (Actual); Study Completion 2018-11-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joanne Filicko-O'Hara, MD, Principal Investigator — Sidney Kimmel Cancer Center at Thomas Jefferson University
Locations (1):
- Thomas Jefferson University, Philadelphia, Pennsylvania, United States

REFERENCES:
- See also: Jefferson University Hospitals — http://www.JeffersonHospital.org

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Bendamustine, Bortezomib, Dexamethasone (Standard)
Started | 24
Completed | 24
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Bendamustine, Bortezomib, Dexamethasone (Standard)
Number analyzed (Participants) | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 18
  >=65 years | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 24
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 14
  White | 10
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 24

OUTCOME MEASURES:

1. Primary Outcome: Count of Participants That Experience Overall Response Following 4 Cycles of the Combination Regimen BBd
Description: ORR (partial remission or better) to induction therapy following 4 cycles of the combination regimen BBd.
Time Frame: At least 140 days
Population: 4 subjects were not evaluable - (1 didn't get any therapy on study, 1 received only first cycle and 2 developed medical issues that took them off study during the first cycle)
Measure: Count of Participants; unit: Participants
Arm/Group | Bendamustine, Bortezomib, Dexamethasone (Standard)
Number analyzed (Participants) | 20
Participants | 13

2. Secondary Outcome: Incidence of Grade 3-4 Adverse Events From the Combination of Bendamustine Hydrochloride, Bortezomib, and Dexamethasone Based on the Common Terminology Criteria Version 4.0
Description: All adverse events are tracked during the course of the trial. Adverse events with a grade of 3-4 will be tracked and recorded.
Time Frame: Up to 1 year
Population: 4 were not evaluable - (1 didn't get any therapy on study, 1 received only first cycle and 2 developed medical issues that took them off study during the first cycle)
Measure: Number; unit: Adverse Events
Arm/Group | Bendamustine, Bortezomib, Dexamethasone (Standard)
Number analyzed (Participants) | 20
Adverse Events | 22

3. Secondary Outcome: Count of Participants That Experience Very Good Partial Remission (VGPR)
Description: Very good partial remission (VGPR) to induction therapy following 4 cycles of the combination regimen BBd. As defined as no dectable M-protein on SPEP (Serum protein electrophoresis) but positive IFX (Immunofixation) on serum or urine and >90% reduction of M-protein in serum and urine
Time Frame: Up to 1 year
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Bendamustine, Bortezomib, Dexamethasone (Standard)
Number analyzed (Participants) | 20
Participants | 9

4. Secondary Outcome: Count of Participants That Experience Progression-free Survival (PFS)
Description: The amount of participants that survive one year after treatment with BBd and do not experience worsening disease.
Time Frame: 1 year
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Bendamustine, Bortezomib, Dexamethasone (Standard)
Number analyzed (Participants) | 20
Participants | 2

5. Secondary Outcome: Count of Participants That Experience Overall Survival (OS)
Description: The amount of participants that start treatment with BBd and survive at least one year post treatment completion.
Time Frame: 1 year
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Bendamustine, Bortezomib, Dexamethasone (Standard)
Number analyzed (Participants) | 20
Participants | 2

ADVERSE EVENTS:
Arm/Group | Bendamustine, Bortezomib, Dexamethasone (Standard)
All-Cause Mortality (participants affected / at risk) | 1/24
Serious Adverse Events (participants affected / at risk) | 9/24
Other Adverse Events (participants affected / at risk) | 24/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bendamustine, Bortezomib, Dexamethasone (Standard) (N=24)
Joint Function Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Death- Anaphylactic Shock (Immune system disorders) | 1 (1)
Hypercalcemia (Blood and lymphatic system disorders) | 1 (1)
Gout (Blood and lymphatic system disorders) | 1 (1)
Syncope episode (Blood and lymphatic system disorders) | 1 (3)
Febrile Neutropenia (Infections and infestations) | 1 (1)
Acute kidney injury (Hepatobiliary disorders) | 1 (2)
Failure to Thrive (General disorders) | 1 (1)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Allergic Reaction (Immune system disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bendamustine, Bortezomib, Dexamethasone (Standard) (N=24)
Alkaline Phosphate increased (Blood and lymphatic system disorders) | 7 (9)
Abdominal cramping (Gastrointestinal disorders) | 1 (1)
Acute kidney injury (Hepatobiliary disorders) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 12 (16)
Anorexia (Psychiatric disorders) | 5 (5)
AST increase (Blood and lymphatic system disorders) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 8 (8)
Bruising (Skin and subcutaneous tissue disorders) | 2 (2)
Change in taste (General disorders) | 4 (4)
Chest pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Confusion (General disorders) | 1 (1)
Conjuctivitis (Eye disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 6 (6)
Creatinine increased (Blood and lymphatic system disorders) | 2 (2)
Decreased Visual Field (Eye disorders) | 1 (1)
Depression (Psychiatric disorders) | 3 (3)
Diarrhea (Gastrointestinal disorders) | 5 (8)
Dry cough (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Dry mouth (General disorders) | 2 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 5 (6)
Edema (General disorders) | 4 (4)
Epistaxis (Blood and lymphatic system disorders) | 1 (1)
Fatigue (General disorders) | 13 (14)
Flu like symptoms (Immune system disorders) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 3 (3)
Hand pain (General disorders) | 1 (1)
Headache (General disorders) | 3 (4)
Hiccups (General disorders) | 1 (2)
Hot flashes (General disorders) | 1 (1)
Hypercalcemia (Blood and lymphatic system disorders) | 4 (4)
Hyperglycemia (Blood and lymphatic system disorders) | 4 (4)
Hyperkalemia (Blood and lymphatic system disorders) | 3 (3)
Hypermagnesemia (Blood and lymphatic system disorders) | 1 (1)
Hypertension (Blood and lymphatic system disorders) | 3 (3)
Hyperuricemia (Blood and lymphatic system disorders) | 3 (3)
Hypoalbuminemia (Blood and lymphatic system disorders) | 3 (3)
Hypocalcemia (Blood and lymphatic system disorders) | 5 (5)
Hypokalemia (Blood and lymphatic system disorders) | 3 (4)
Hypomagnesium (Blood and lymphatic system disorders) | 2 (2)
Hyponatremia (Blood and lymphatic system disorders) | 3 (3)
Hypophosphatemia (Blood and lymphatic system disorders) | 4 (5)
Hypotension (Blood and lymphatic system disorders) | 2 (2)
Infection site reaction (Infections and infestations) | 4 (4)
Insomnia (General disorders) | 3 (3)
Leg Pain (spasm) (Musculoskeletal and connective tissue disorders) | 1 (1)
Light headedness (General disorders) | 1 (1)
Loss of appetite (General disorders) | 2 (2)
Lymphocyte count decreased (Blood and lymphatic system disorders) | 6 (15)
Nasal Congestion (General disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 9 (10)
Neuropathy (Nervous system disorders) | 2 (2)
Orthostatic hypotension (Blood and lymphatic system disorders) | 1 (1)
Pain (General disorders) | 3 (4)
Pain at port site (General disorders) | 1 (1)
Pain Knee (General disorders) | 1 (2)
Pain shoulder (General disorders) | 1 (1)
Pain- side of face (General disorders) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1)
Paresthesia (Nervous system disorders) | 1 (1)
peripheral motor neuropathy (Nervous system disorders) | 1 (1)
Platelet Count decreased (Blood and lymphatic system disorders) | 2 (3)
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rash unspecified (Skin and subcutaneous tissue disorders) | 1 (1)
Rib pain (General disorders) | 2 (2)
Sinusitis (Infections and infestations) | 1 (2)
Sore Throat (General disorders) | 2 (2)
Soreness (General disorders) | 1 (2)
Stomach Pain (Gastrointestinal disorders) | 1 (1)
Urinary Frequency (Renal and urinary disorders) | 2 (2)
Weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
White blood cell count decreased (Blood and lymphatic system disorders) | 7 (14)
Swelling L- Breast (Reproductive system and breast disorders) | 1 (1)
Urinary Tract infection (Renal and urinary disorders) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Indigestion (Gastrointestinal disorders) | 1 (1)
Hematuria (Renal and urinary disorders) | 2 (2)
Gum infection (Infections and infestations) | 1 (1)
Fall (General disorders) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Ear infection (Ear and labyrinth disorders) | 1 (2)
ANC increased (Blood and lymphatic system disorders) | 1 (1)
Allergic Rhinitis (General disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes